CLINICAL TRIAL: NCT00242398
Title: Heparin Free Hemodialysis for Patients With Bleeding High Risk in ICU. Randomized Study: Heparin Free Dialysis With Intermittent Saline Flushes Versus Heparin Free Dialysis With Nephral 400ST (AN69ST, Hospal, France)
Brief Title: Hemodialysis Without Anticoagulation in Intensive Care Unit
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Départemental (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HDI-FH
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-10

CONDITIONS: Kidney Failure; Critically Ill; Hemorrhage
Keywords: Intensive care unit; Patients with bleeding high risk; Intermittent hemodialysis without anticoagulation; Blood lost
MeSH Terms: conditions — Renal Insufficiency; Critical Illness; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AN69 ST

SUMMARY:
The purpose of this study is to determine the safety and operative efficacy of intermittent hemodialysis without anticoagulation with saline flushes or Nephral 400ST in patients at high risk of bleeding

DETAILED DESCRIPTION:
Hemodialysis in patients who are at high risk of bleeding complications represents a challenge of balancing the needs for establishment of an adequately functioning extracorporeal circuit for dialytic therapy with the requirement of not exacerbating existing bleeding or precipitating bleeding in predisposed subjects.

Several methods of nonheparin dialysis have been used. The method most commonly used to effect such treatment is "saline flushing": saline boluses are delivred at frequent intervals. This method is far from optimal for several reasons, including failure to maintain a patent circuit in significant proportion of patients, an added logistic burden on dialysis nurses. An alternative method of avoiding systemic heparinization is priming the dialysis membrane with heparin before hemodialysis. The method is based on fact that AN69ST (Nephral 400ST , Hospal, France) dialysis membrane have a high affinity for binding heparin, and that the bound heparin exerts a localized antithrombotic effect without systemic spillover.

Comparison: heparin free hemodialysis with saline flushes compared heparin free hemodialysis with Nephral 400ST.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patient with high risk bleeding
* patient requiring dialytic therapy in intensive care unit

Exclusion Criteria:

* Pregnancy
* History of heparin-induced thrombocytopenia or serious heparin allergy
* History of serious membrane dialysis allergy
* Treatment by any of following medications 24H within the inclusion:

prophylactic or therapeutic anticoagulation with unfractioned heparin or low molecular weight heparin nonsteroidal anti-inflammatory agents direct thrombin inhibitors, antithrombin concentrate, activated protein C, anti-factor Xa pentasaccharide

* Treatement by acetylsalicylic acid or other antiplatelet agent excluding platelet glycoprotein IIb/IIIa antagonists 7 days within the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-10; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Early stop dialysis treatment for rapid and persistent elevations in venous extracorporeal pressure secondary to extracorporeal thrombosis. | at the end of the dialysis treatement

SECONDARY OUTCOMES:
Blood lost associated with extracorporeal thrombosis or active bleeding | At the end of the dialysis treatment
Necessary time of nurse's work | During the dialysis treatment
Weight lost patients during dialysis treatment | At the end of dialysis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Martin-Lefèvre, Principal Investigator
Locations (1):
- CHD, La Roche-sur-Yon, France